CLINICAL TRIAL: NCT03620045
Title: An Exercise Intervention to Improve the Eating Patterns of Preadolescent Children
Brief Title: An Exercise Intervention to Improve the Eating Patterns of Preadolescent Children at High Risk for Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Responsible Party: Principal Investigator, Nichole Kelly, Associate Professor, University of Oregon
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 04252017.043
Record Dates: First submitted 2018-07-27; First posted 2018-08-08 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Eating Behavior; Self-Regulation
MeSH Terms: conditions — Feeding Behavior; Self-Control

STUDY DESIGN:
Intervention Model Description: Randomized crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute moderate physical activity (Experimental): Participants will walk at a moderate intensity for 20 minutes on a treadmill
  Interventions: Behavioral: Acute moderate physical activity
- Sedentary activity (No Intervention): Participants will be permitted to read books and/or draw for 20 minutes

INTERVENTIONS:
Behavioral: Acute moderate physical activity — For 20 minutes, participants will walk on a treadmill at a moderate intensity based on a combination of evidence-based and pre-determined parameters, including ratings of perceived exertion and heart rate
  Arms: Acute moderate physical activity

SUMMARY:
Children in rural communities experience significant obesity-related health disparities; they are 26%-55% more likely to be obese and less likely to have health insurance and access to weight management specialists than are their urban peers. Geographic-specific disparities in obesity may be due, in part, to variations in eating behaviors. Children in rural communities describe purchasing and consuming significantly more energy-dense, low-nutrient food items relative to their urban peers. Existing behavioral strategies for improving children's EI patterns have largely been ineffective in reducing risk for excess weight gain. The primary aim of the proposed study is to test the effects of a brief, novel strategy for improving rural children's eating behaviors. Specifically, the study aims to harness the well-documented benefits of an acute bout (20 min) of moderate physical exercise on children's executive functioning, and to see if these cognitive changes lead to better self-regulation of eating. If 20 min of moderate physical exercise is associated with observed improvements in preadolescent children's eating secondary to increases in executive functioning, these data may offer explicit targets for an obesity prevention trial in rural Oregon elementary schools.

ELIGIBILITY:
Inclusion criteria:

* 8-10 years (block recruited to ensure 50% female, 50% obese)
* Rural geographic location (≥ 10 miles from a city of ≥ 40,000)
* Understand English

Exclusion criteria

* BMI < 5th percentile
* Major medical condition, current full-threshold psychiatric diagnosis, or moderate suicide risk (e.g., plan or intent)
* Current or recent use (< 3 months) of medication known to affect body weight or energy intake
* Recent brain injuries that would be expected to affect neuropsychological functioning
* Mobility impairments that would impede their ability to walk on a treadmill
* Estimated full-scale intelligence quotient score ≤ 70
* History of pregnancy
* Significant food allergies that would prevent them from safely consuming the study's breakfast and lunch meals
* Responses on a food preference questionnaire that suggest that they do not like (i.e., rated them below 6 on a scale from 1 to 10) at least 50% of the food items offered in the lunch test meal

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — We do not confirm sex based on any biological testing; as such, we will rely on self- and parent-reported gender identity for each participating child; we have no exclusion criteria based on gender
Enrollment: 92 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2021-08-04 (Actual)

PRIMARY OUTCOMES:
Energy intake | up to 14 days
  total kcal consumed during a laboratory test meal after each of two conditions

SECONDARY OUTCOMES:
Executive functioning | Assessed immediately after each of the two experimental conditions administered during two separate study visits approximately 14 days of each other
  executive functioning performance assessed with a 3-minute task immediately after each of two conditions

CONTACTS AND LOCATIONS:
Overall Officials: Nichole R Kelly, PhD, Principal Investigator — University of Oregon
Locations (1):
- University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kelly NR, Guidinger C, Swan DM, Thivel D, Folger A, Luther GM, Hahn ME. A brief bout of moderate intensity physical activity improves preadolescent children's behavioral inhibition but does not change their energy intake. J Behav Med. 2024 Aug;47(4):692-706. doi: 10.1007/s10865-024-00495-1. Epub 2024 Apr 26. PMID 38671287